CLINICAL TRIAL: NCT04816968
Title: TAID Study - A Prospective Interventional Trial on Antibiotics Continuous Infusion at Home
Brief Title: Antibiotics Continuous Infusion at Home
Acronym: TAID
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ospedale San Carlo Borromeo (Other)
Collaborators: Associazione Oncologica Milanese AmoLaVita ONLUS (Unknown)
Responsible Party: Principal Investigator, Vittorio Montefusco, Medical Director Ssd of Oncohematology, Ospedale San Carlo Borromeo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAID Study
Record Dates: First submitted 2021-03-22; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Severe Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — Cefepime; Piperacillin, Tazobactam Drug Combination; Meropenem; Vancomycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A - Cefepime (Experimental): Continuous infusion of Cefepime at home.
  Interventions: Drug: Cefepime
- Arm B - Piperacillin/tazobactam (Experimental): Continuous infusion of Piperacillin/tazobactam at home.
  Interventions: Drug: Piperacillin/tazobactam
- Arm C - Meropenem (Experimental): Continuous infusion of meropenem at home.
  Interventions: Drug: Meropenem
- Arm D - Vancomycin (Experimental): Continuous infusion of vancomycin at home.
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Cefepime — Cefepime from 3 to 6 gr, based on patient's clinical status, reduced dose based on organ function and physician discretion, in 100cc saline solution in elastomer, perfused in 24 hours.
  Arms: Arm A - Cefepime
Drug: Piperacillin/tazobactam — Piperacillin/Tazobactam 18 gr, based on patient's clinical status, reduced dose based on organ function and physician discretion, in 100cc saline solution in elastomer, perfused in 24 hours.
  Arms: Arm B - Piperacillin/tazobactam
Drug: Meropenem — Meropenem 3 gr, based on patient's clinical status, reduced dose based on organ function and physician discretion, in 100cc saline solution in elastomer, perfused in 24 hours.
  Arms: Arm C - Meropenem
Drug: Vancomycin — Vancomycin 30 mg/kg, based on patient's clinical status, reduced dose based on organ function and physician discretion, in 100cc saline solution in elastomer, perfused in 24 hours.
  Arms: Arm D - Vancomycin

SUMMARY:
BACKGROUND: The spread of multidrug-resistant bacteria represents a well-known problem, which must be face up by optimizing antibiotic therapy both in terms of choosing the most appropriate drug and of an adequate treatment duration. The method of administration is also a critical element. There are data relating to the maximization of the efficacy of Carbapenems and Piperacillin/Tazobactam by continuous infusion, able to constantly maintain adequate drug concentrations. Several studies, conducted comparing a standard administration of Carbapenem or Piperacillin/Tazobactam to an extended administration or continuous perfusion to evaluate safety and efficacy in terms of mortality reduction, have been documented. The achievement of optimal serum concentrations during continuous infusion has been documented both for Carbapenems and Piperacillin/Tazobactam, and for other types of antibiotics such as Cefepime and Vancomycin. The duration of antibiotic treatment is a critical factor for the prevention of relapses as well as the onset of resistance. The recommended duration of antibiotic treatment varies according to the site of infection and the type of pathogen and is generally between 7 and 14 days, however, in particular cases it is possible that the administration of antibiotics must be longer than one month. In general, the length of hospitalization is associated with a greater likelihood of complications for patients, with a substantial increase in the risk of developing multiple types of complications, such nosocomial infections, bed rest, bedsores, falls, malnutrition and disorientation. It should also be noted that prolonged hospitalization leads to a substantial increase in care costs. The advantage in terms of greater therapeutic success linked to the continuous infusion of some types of antibiotics has been used for the development of home infusion protocols for antibiotic therapy. There are numerous studies that show the feasibility and effectiveness of home infusion antibiotic therapy using elastomeric devices, documenting its substantial equivalence with respect to hospital treatment. The antibiotics for which there is evidence of feasibility are various, including Cefepime, Vancomycin and Piperacillin/Tazobactam.

STUDY DESIGN: The study is aimed to patients with severe bacterial infections who have started an antibiotic treatment and are benefiting from such therapy. The purpose of the study is to move the continuation of antibiotic therapy to the home setting once its efficacy and tolerability during hospitalization have been documented, in order to allow the patient a potentially eradicating treatment, of adequate duration without the need of hospitalization. Patients are enrolled when the efficacy and tolerability of the ongoing antibiotic treatment based on Cefepime, Meropenem, Piperacillin/Tazobactam or Vancomycin has been documented. The protocol requires that the patient go to the hospital every morning to replace the elastomer and to carry out a medical examination. Blood chemistry tests, which include at least blood counts, electrolytes, renal function, liver function and inflammation indices are scheduled to be performed at least once a week. Exams can also be done more frequently based on clinical needs. Antibiotic therapy should be carried out until the infection is cured, as per current clinical practice. For the purposes of the study, the patient remains under observation for 30 days after enrollment. Blood samples for the assessment of antibiotic concentrations will be performed in correspondence with the blood chemistry tests performed routinely for patient assessment. In any case, for each patient, a sample is taken for the dosage of the antibiotic used, which will be a single sample in the event of a continuous infusion, or a downstream sample (within one hour of the new antibiotic administration) and peak (30 minutes after the end of the infusion). The pharmacokinetic sampling relating to the outpatient phase will be carried out on the third or fourth day of continuous infusion therapy at the time of the elastomer change.

DETAILED DESCRIPTION:
STATISTICAL ANALYSIS: This is an interventional monocentric study. The primary endpoint of the study is a reduction in hospitalization days. The study population is divided into 4 treatment arms: assuming that the average length of hospitalization for the standard treatment of a severe infection, for each of the types of antibiotic studied, is 14 days, with the treatment envisaged by the study it is assumed to reduce this duration,for all 4 treatment arms, to a number equal to or less than 12 days. With these premises, applying the One sample t-test design method, assuming α = 0.05 and β = 0.1, the number of patients expected is 9 for each treatment arm. Considering a 30% dropout, the total population to be enrolled for each type of antibiotic is 12 patients. In total, the study will enroll 48 patients. The study provides for an observation period of 30 days from enrollment. During this period, efficacy, safety and pharmacokinetic data will be collected for each treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 90 years.
* Ability to understand and sign informed consent.
* Treatment infection responsive to Cefepime, Meropenem or Piperacillin / Tazobactam, Vancomycin.
* Absence of allergies to Cefepime, Meropenem or Piperacillin / Tazobactam, Vancomycin.
* Evidence of clinical response to treatment with Cefepime, Meropenem or Piperacillin / Tazobactam, Vancomycin and at least 3 days of apyrexia with current infusion antibiotic therapy.
* Good tolerance to ongoing antibiotic treatment with Cefepime, Meropenem or Piperacillin / Tazobactam, Vancomycin.

Exclusion Criteria:

* Inability for any reason (e.g. absence of caregiver) to manage the elastomeric pump and access the hospital on a daily basis.
* Lack of adequate venous access.
* Inability to hydrate themselves properly orally.
* Infection involving the central nervous system.
* Creatinine> 2 mg / dL.
* Neutrophil granulocytes ≤ 1000 / µL.
* Platelets ≤ 20000 / µL.
* "aspartate amino transferase" and "alanine amino transferase" > 100 U / L.
* Bilirubin> 3 mg / dL.
* Presence of any comorbidities that, in the opinion of the physician, could compromise the safe execution of antibiotic home continuous infusion.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of hospitalization days for the treatment of severe bacterial infections | 14 days
  The number of hospitalization days for the treatment of severe bacterial infections with continuous infusion antibiotics at home will be compared with the number of hospitalization days for standard antibiotics therapies for severe bacterial infections.

SECONDARY OUTCOMES:
Effectiveness of antibiotic treatment | 30 days from the enrollment
  The effectiveness of antibiotic treatment in continuous infusion at home will be compared with the effectiveness of antibiotic standard treatment in terms of the number of patients that have to start a new antibiotic line therapy.
Number of new hospitalizations days for the same problem in the month following the start of home continuous infusion therapy. | 30 days from the enrollment
  The number of new hospitalizations days for the same problem in the month following the start of continuous infusion antibiotic therapy at home will be compared with the number of new hospitalizations for the same problem with antibiotic standard treatment.
Ongoing adverse events of home continuos infusion therapy. | 30 days from the enrollment
  The number of adverse events of each grade will be quantified.
Adverse events related to the presence of a venous access | 30 days from the enrollment
  The number of adverse events related to the presence of a venous access will be quantified.

CONTACTS AND LOCATIONS:
Overall Officials: Vittorio Motefusco, MD, Principal Investigator — Ospedale San Carlo Borromeo
Locations (1):
- ASST Santi Paolo Carlo - San Carlo Borromeo Hospital - SSd Onco-Hematology, Milan, Italy

REFERENCES:
- [Background] Falagas ME, Tansarli GS, Ikawa K, Vardakas KZ. Clinical outcomes with extended or continuous versus short-term intravenous infusion of carbapenems and piperacillin/tazobactam: a systematic review and meta-analysis. Clin Infect Dis. 2013 Jan;56(2):272-82. doi: 10.1093/cid/cis857. Epub 2012 Oct 16. PMID 23074314
- [Background] Grant EM, Kuti JL, Nicolau DP, Nightingale C, Quintiliani R. Clinical efficacy and pharmacoeconomics of a continuous-infusion piperacillin-tazobactam program in a large community teaching hospital. Pharmacotherapy. 2002 Apr;22(4):471-83. doi: 10.1592/phco.22.7.471.33665. PMID 11939682
- [Background] Lau WK, Mercer D, Itani KM, Nicolau DP, Kuti JL, Mansfield D, Dana A. Randomized, open-label, comparative study of piperacillin-tazobactam administered by continuous infusion versus intermittent infusion for treatment of hospitalized patients with complicated intra-abdominal infection. Antimicrob Agents Chemother. 2006 Nov;50(11):3556-61. doi: 10.1128/AAC.00329-06. Epub 2006 Aug 28. PMID 16940077
- [Background] Lodise TP Jr, Lomaestro B, Drusano GL. Piperacillin-tazobactam for Pseudomonas aeruginosa infection: clinical implications of an extended-infusion dosing strategy. Clin Infect Dis. 2007 Feb 1;44(3):357-63. doi: 10.1086/510590. Epub 2007 Jan 2. PMID 17205441
- [Background] Voumard R, Gardiol C, Andre P, Arensdorff L, Cochet C, Boillat-Blanco N, Decosterd L, Buclin T, de Valliere S. Efficacy and safety of continuous infusions with elastomeric pumps for outpatient parenteral antimicrobial therapy (OPAT): an observational study. J Antimicrob Chemother. 2018 Sep 1;73(9):2540-2545. doi: 10.1093/jac/dky224. PMID 29982449
- [Background] Care of the elderly patient. J. Hosp. Med 2006;1;60-61
- [Background] Lagoe RJ, Johnson PE, Murphy MP. Inpatient hospital complications and lengths of stay: a short report. BMC Res Notes. 2011 May 5;4:135. doi: 10.1186/1756-0500-4-135. PMID 21545741
- [Background] Hoogervorst-Schilp J, Langelaan M, Spreeuwenberg P, de Bruijne MC, Wagner C. Excess length of stay and economic consequences of adverse events in Dutch hospital patients. BMC Health Serv Res. 2015 Dec 1;15:531. doi: 10.1186/s12913-015-1205-5. PMID 26626729
- [Background] Manning L, Wright C, Ingram PR, Whitmore TJ, Heath CH, Manson I, Page-Sharp M, Salman S, Dyer J, Davis TM. Continuous infusions of meropenem in ambulatory care: clinical efficacy, safety and stability. PLoS One. 2014 Jul 14;9(7):e102023. doi: 10.1371/journal.pone.0102023. eCollection 2014. PMID 25019523